CLINICAL TRIAL: NCT04017000
Title: BLAdder Shape Test: Medium-fill Cystometry and Trans-abdominal Assessment of Bladder Shape in Women With Overactive Bladder
Brief Title: Bladder Shaper Test
Acronym: BlaST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: STH20318
Record Dates: First submitted 2019-07-02; First posted 2019-07-12 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Diagnosis of Urinary Tract Symptons

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinician performing patient Urodynamics will be different from the clinician who undertakes the bladder shape test.
  Urodynamics clinician will be blinded to the results of the bladder shape test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BlaST study (Active Comparator): Patients scheduled for Urodynamic clinic will be offered to participate in the study. Once consented to participate, the participant will be scheduled for a bladder shape test clinic at least one week in advance of their Urodynamic appointment. At their blast clinic, participants will attend a clinical room with a portable bladder scanner. Participants will be asked to consume up to 1000 mls of water over a 20-30 period until their bladder is full. The participant will have their bladder scanned at 10 minute intervals during the filling phase and after prompted voiding.
  The participants Urodynamic clinic will run according to routine care.
  Interventions: Diagnostic Test: Bladder Shape Test
- Calibration Sub Study (Other): Any patients who are not eligible or decline participation in the main study will be offered the chance to participate in the calibration sub study.
  Participants will be scheduled for their clinically indicated Urodynamic appointment where they will have their bladder imaged by portable ultrasound.
  Participants will consent for these images to be used as part of the calibration of the technology being used to measure bladder shape change.
  Interventions: Other: Calibration images

INTERVENTIONS:
Diagnostic Test: Bladder Shape Test — Capturing images of bladder under natural filling conditions images are analysed at a later date for shape change.
  Arms: BlaST study
Other: Calibration images — Capturing images of bladder under artificial filling conditions during Urodynamic assessment images are analysed at a later date to inform shape change technology.
  Arms: Calibration Sub Study

SUMMARY:
This study is comparing a novel method of Bladder shape measurements using ultrasound for diagnosis of lower urinary tract symptoms in comparison to traditional Urodynamic assessment. All participants will undergo the novel investigation followed by their usual Urodynamics.

DETAILED DESCRIPTION:
This study hypothesises that bladder shape changes associated with involuntary contractions of the detrusor muscle, might be detected using trans abdominal ultrasound, which could itself form the basis of a novel diagnostic test for detecting involuntary contractions associated with overactive bladder syndrome and urgency incontinence.

The detection of involuntary bladder contractions currently relies on invasive internal pressure measurement, commonly termed Urodynamics. This is an invasive test involving the placement of pressure measurement catheters, usually via the urethra into the bladder and via the anal canal into the rectum. In its normal healthy state, the bladder remains a contractile throughout filling and is compliant, meaning that there is minimal or zero increase in pressure as it fills. During Urodynamics, the bladder is filled artificially, using a pump, with water or contrast medium via a urethral catheter, whilst abdominal pressure is measured via a rectal catheter introduced anally. Differences between pressure measurements in the bladder and the abdomen are used to detect involuntary detrusor contractions; termed 'detrusor over activity when detected during Urodynamics. Patients often report Urodynamics as being uncomfortable and undignified, and the test carries a risk of introducing urinary tract infection. Furthermore, there are significant issues relating to the sensitivity of Urodynamics in the detection of abnormal bladder contractions in the context of Overactive Bladder.

Variations in bladder shape have been observed in association with detrusor over activity during video-Urodynamics, when fluoroscopic images are captured during filling with contrast medium. At one extreme, women with neuropathic overactive bladder have been observed to have tense, spherical or dome-shaped bladders with trabeculations 'fir tree' or 'Christmas tree' bladder. In women with normal detrusor muscle function, the bladder outline appears relaxed and a contractile, following the contours of the pelvis when assessed by cystography.

Although conventional Urodynamics has previously been regarded as the 'Gold Standard' in the assessment of lower urinary tract disorders, it is also well recognised as having issues of sensitivity, patient acceptability and cost. The test is commonly employed to diagnose and better understand the underlying pathophysiology of incontinence and is often deemed necessary, particularly prior to invasive forms of treatment. The requirement for urodynamic equipment, including its purchase, maintenance, associated training and size restricts its use to specialist hospital facilities, rendering it relatively inaccessible as a diagnostic tool. In addition to this patients have reported finding Urodynamics embarrassing and uncomfortable and with the inclusion of x-ray screening (video-cystometry) which is part of the procedure which aims to contemporaneously evaluate lower urinary tract structure and morphology, involves exposure to ionising radiation and is of unproven benefit. Therefore, there is a patient & clinical need to objectively assess lower urinary tract function with less invasive, sensitive, reproducible and more widely available tests.

A pilot study will now be performed to establish the use of bladder shape testing as a new investigation for the assessment and diagnosis of lower urinary tract disorders. It is anticipated that this pilot will lead to the development of a new healthcare product that can be used in the primary care setting as an alternative to urodynamic assessment in the acute secondary care environment.

ELIGIBILITY:
Inclusion Criteria:

* Women referred for urodynamic evaluation of LUTS, including urinary storage symptoms, with or without incontinence.
* Women aged 18 years and over.
* Women willing and able to discontinue any current anticholinergic medication for a minimum period of 10 days prior to starting any study-related procedure.
* Women who understand and are willing and feel able to comply with the study protocol/procedures and who have provided written informed consent.

Exclusion Criteria:

* Current pregnancy
* Suspicion of pelvic malignancy
* Unable to consume 1000ml still water over 20 minutes
* Current urinary tract infection (UTI) (as assessed by urine dipstick and symptomatology. Patients with current UTI will be treated and further BlaST/Urodynamics appointments offered as appropriate. Women with cyclical urinary symptoms in association with menstrual cycle will be scheduled for BlaST and conventional Urodynamics at the same time each month, other patients will receive both tests usually within a month of each other, but never on the same day.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study only available to women attending Urogynaecology clinics
Enrollment: 156 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Recruitment | At 12 months
  Assessing recruitment rate for a larger study
Participants Completion Rate | At 12 months
  Assessing drop out and completing patients to inform sample size for larger study

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Radley, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No